CLINICAL TRIAL: NCT04763837
Title: Migration of Intraureteral Stents Compared to Conventional Double-J Stents.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to continue
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Kellen Choi, Asst Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20.0563
Record Dates: First submitted 2021-01-28; First posted 2021-02-21 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Urologic Diseases; Urological System Complication of Procedure
Keywords: urology; ureteral stent
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, randomized controlled, single-blinded trial. The subjects will include up to 140 patients (about 70 subjects per group) from ages 1-100 years old that are to undergo stent placement for nephrolithiasis, hydronephrosis, and urological cancer. They will be randomized to one of two groups: intraureteral stent or conventional double-J stent. Upon removal of the stent, migration distance will be measured via fluoroscopy using a calibrated x-ray system.
Who Masked: Participant
Masking Description: Subjects will not be informed of which type of ureteral stent will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intraureteral stent group (Experimental): Patients assigned to this group will undergo placement of an intraureteral stent, a tube that drains urine from the kidney to the bladder and has a loop of tube in only in the kidney and NOT in the bladder. This group will be the experimental group.
  Interventions: Device: Intraureteral stent
- Conventional Double-J stent (Active Comparator): Patients assigned to this group will undergo placement of a double-J ureteral stent, a tube that drains urine from the kidney to the bladder and has a loop of tube in both the kidney and the bladder. This group will serve as the control.
  Interventions: Device: Conventional Double-J stent

INTERVENTIONS:
Device: Intraureteral stent — This intervention involves the placement of an intraureteral stent, a tube that drains urine from the kidney to the bladder and has a loop of tube only in the kidney and NOT in the bladder. The distal end of the tube will stay in the ureter just proximal to the opening to the bladder.
  Other Names: Polaris™ Loop Ureteral Stent - Boston Scientific
  Arms: Intraureteral stent group
Device: Conventional Double-J stent — This intervention involves the placement of a conventional double-J stent, a tube that drains urine from the kidney to the bladder and has a loop of tube in both the kidney and in the bladder.
  Arms: Conventional Double-J stent

SUMMARY:
The purpose of this study is to determine if stents placed with only one loop in the kidney move more than stents placed with a loop in both the kidney and a bladder. Participants in this study will undergo placement of a stent into the ureter that drains urine from the kidney into the bladder. The stent will be placed in 1 of 2 ways: either with only a loop of the stent is left in the kidney or in the regular manner where a loop of the stent is left in both the kidney and in the bladder. The position of the stent will be measured at the time of placement. When the stent is removed, the position of the stent will be measured prior to pulling the stent.

DETAILED DESCRIPTION:
The ureteral stent is one of the most extensively used tools in the field of urology. They are used for aiding post-operative healing of the ureter, visualizing the ureteral during procedures, and alleviating ureteral obstruction (eg. nephrolithiasis). Double-J stents, which are secured by loops in both the renal pelvis and the bladder, have become most urologists' go-to choice for ureteral stents since they were introduced in the 1970s. Unfortunately, it has been shown that 80-90% of patients with ureteral stents have urinary complaints following stent placement.

Interestingly, a recent study suggested utility of intraureteral stents. These stents have one loop in the renal pelvis while their distal end is positioned proximal to the ureteral orifice. The above-mentioned study showed that patients with intraureteral stents had less discomfort as opposed to the those that had double-J stents.

Due to the immense number of patients that require ureteral stent placement, this improvement in comfort is very promising for the urological field. However, no one has studied if stents placed intraureterally migrate from the time they are placed to the time they are removed. If stents migrate proximally toward the renal pelvis, it is possible that retrieval could be more difficult, and the ureteral patency established by the stent could be compromised.

The objective of this study is to determine if intraureterally placed stents migrate as compared to ureteral stents placed via the conventional method.

This study will be a prospective, randomized controlled, single-blinded trial. The subjects will include up to 140 patients (about 70 subjects per group) from ages 1-100 years old that are to undergo stent placement for nephrolithiasis, hydronephrosis, and urological cancer.

Prior to the procedure, each patient that has agreed to participate in this study will be randomly assigned to receive a stent placed intraureterally or a stent placed in the conventional manner. After each intraureteral stent is placed via cystoscopy, the distance of the distal end of the stent to the ureteral orifice will be measured via fluoroscopy that was calibrated prior to the procedure. After each double-J stent is placed via cystoscopy, the length of stent that is present in the bladder will also be measured using calibrated fluoroscopy . Subjects will not be informed of which group they are assigned to. When the patients return for stent removal, the previously mentioned distances will be measured again prior to pulling the stent. They will also be asked to complete the ureteral stent symptom questionnaire (USSQ) to assess stent-associated discomfort. The primary endpoint of the study would be stent migration distance (mm). Secondary endpoints would include patient comfort level.

All medical records will be accessed on secure devices and networks. All subjects will be assigned a subject number upon enrolled in the study. When a researcher needs to record data from a patient's medical records, they will record this information with the patient's corresponding subject number. Only the researchers involved in this study will have access to the document that includes patient identifiers and their subject number. At the conclusion of this study, the document with patient identifiers and subject numbers will be destroyed.

Data will be collected from electronic medical records of patients from ULP (University of Louisville Physicians) Urology.

ELIGIBILITY:
Inclusion Criteria:

* Those undergoing ureteral stent placement for nephrolithiasis, hydronephrosis, and urological cancer.

Exclusion Criteria:

* none

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-02 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Stent migration | 12 months
  The distance that the stent migrates into the bladder or into the kidney.

SECONDARY OUTCOMES:
Patient comfort level | 12 months
  Patient comfort level, as assessed via the Ureteral stent symptom questionnaire (USSQ).

CONTACTS AND LOCATIONS:
Overall Officials: Kellen B Choi, DO, FACOS, Principal Investigator — Associate Professor, University of Louisville Department of Urology

REFERENCES:
- [Background] Finney RP. Experience with new double J ureteral catheter stent. 1978. J Urol. 2002 Feb;167(2 Pt 2):1135-8; discussion 1139. doi: 10.1016/s0022-5347(02)80361-5. No abstract available. PMID 11905888
- [Background] Joshi HB, Okeke A, Newns N, Keeley FX Jr, Timoney AG. Characterization of urinary symptoms in patients with ureteral stents. Urology. 2002 Apr;59(4):511-6. doi: 10.1016/s0090-4295(01)01644-2. PMID 11927301
- [Background] Pollard SG, Macfarlane R. Symptoms arising from Double-J ureteral stents. J Urol. 1988 Jan;139(1):37-8. doi: 10.1016/s0022-5347(17)42282-8. PMID 2961892
- [Background] Yoshida T, Inoue T, Taguchi M, Matsuzaki T, Murota T, Kinoshita H, Matsuda T. Efficacy and Safety of Complete Intraureteral Stent Placement versus Conventional Stent Placement in Relieving Ureteral Stent Related Symptoms: A Randomized, Prospective, Single Blind, Multicenter Clinical Trial. J Urol. 2019 Jul;202(1):164-170. doi: 10.1097/JU.0000000000000196. Epub 2019 Jun 7. PMID 30829132
- [Background] Joshi HB, Newns N, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG. Ureteral stent symptom questionnaire: development and validation of a multidimensional quality of life measure. J Urol. 2003 Mar;169(3):1060-4. doi: 10.1097/01.ju.0000049198.53424.1d. PMID 12576846